CLINICAL TRIAL: NCT00397046
Title: An Ascending and Multiple Dose Study of the Safety, Tolerability, and Pharmacokinetics of HKI-272 Administered Orally to Japanese Subjects With Advanced Solid Tumors
Brief Title: A Study Of The Safety And Tolerability Of HKI-272 Administered Orally To Japanese Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-104
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Tumors
Keywords: Advanced Malignant Solid Tumors; HKI-272; Neratinib; Nerlynx
MeSH Terms: conditions — Neoplasms | interventions — neratinib

STUDY DESIGN:
Intervention Model Description: This was an open-label, phase 1, ascending single and multiple oral dose study of neratinib administered to subjects with advanced solid tumors. Each subject participated in only 1 dose group and received a single dose of neratinib. This was followed by a 1-week observation period, and the subject then received neratinib administered as a continual oral daily dose for up to 6 months (6 cycles). Daily dose administration could continue beyond 6 cycles at the same dose level after consultation with the sponsor if neratinib was well tolerated and there was no evidence of progressive disease.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Neratinib 80 mg (Experimental)
  Interventions: Drug: neratinib
- Neratinib 160 mg (Experimental)
  Interventions: Drug: neratinib
- Neratinib 240 mg (Experimental)
  Interventions: Drug: neratinib
- Neratinib 320 mg (Experimental)
  Interventions: Drug: neratinib

INTERVENTIONS:
Drug: neratinib — HKI-272

SUMMARY:
The purpose of this study is to assess the tolerability and safety of HKI-272, and to determine the maximum dose that can safety be given. The secondary purpose of this study is to determine how the body uses and gets rid of HKI-272 and to assess whether HKI-272 is effective for the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase 1 open-label sequential-group study of ascending single and multiple oral doses administered to subjects with advanced solid tumors. Each subject will participate in only 1 dose group and will receive a single dose of test article, followed by a 1-week observation period, and then will receive the test article administered once-daily by mouth in cycles consisting of 28 days. Subjects will be enrolled in groups of 3 to 6. Adverse events and dose-limiting toxicities will be assessed from the first single dose.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of metastatic or advanced cancer that has failed standard effective therapy
2. Life expectancy of at least 12 weeks and adequate performance status
3. Adequate bone marrow, kidney and liver function
4. Willingness of male and female subjects who are not surgically sterile or post-menopausal to use adequate methods of birth control

Exclusion Criteria

1. Any anticancer chemotherapy, radiotherapy immunotherapy or investigational agents within 4 weeks of first dose of HKI-272
2. Inadequate cardiac function
3. Surgery within 2 weeks of first dose of HKI-272
4. Active central nervous system metastases (i.e., symptomatic, required use of corticosteroids and/or progressive growth)
5. Significant gastrointestinal disorder with diarrhea as a major symptom
6. Pregnant or breast feeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (2):
- Japan (2):
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto, Tokyo
  - Shizuoka Cancer Center, Shizuoka

REFERENCES:
- [Derived] Ito Y, Suenaga M, Hatake K, Takahashi S, Yokoyama M, Onozawa Y, Yamazaki K, Hironaka S, Hashigami K, Hasegawa H, Takenaka N, Boku N. Safety, efficacy and pharmacokinetics of neratinib (HKI-272) in Japanese patients with advanced solid tumors: a Phase 1 dose-escalation study. Jpn J Clin Oncol. 2012 Apr;42(4):278-86. doi: 10.1093/jjco/hys012. Epub 2012 Feb 27. PMID 22371427

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib 80 mg: Neratinib 80 mg qd
- Neratinib 160 mg: Neratinib 160 mg qd
- Neratinib 240 mg: Neratinib 240 mg qd
- Neratinib 320 mg: Neratinib 320 mg qd
Period: Overall Study
Arm/Group | Neratinib 80 mg | Neratinib 160 mg | Neratinib 240 mg | Neratinib 320 mg
Started | 3 | 3 | 10 | 5
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 10 | 5
Not completed — Disease Progression | 3 | 3 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib 80 mg | Neratinib 160 mg | Neratinib 240 mg | Neratinib 320 mg | Total
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 3 | 14
  >=65 years | 0 | 0 | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.67 (9.50) | 48.33 (5.13) | 62.50 (10.19) | 59.40 (7.64) | 58.48 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 8
  Male | 2 | 1 | 8 | 2 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 3 | 3 | 10 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: DLT was defined as any drug-related nonhematologic grade 3 or any grade 4 adverse event (AE) according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0, except the grade 3 nausea, vomiting, diarrhea, or rash, unless the subject was receiving appropriate medical therapy. Additional DLTs included the following: grade 2 or 3 diarrhea lasting 2 or more days for which the subject was receiving medical therapy or that was associated with fever or dehydration.
Time Frame: First dose date through 21 days
Population: All subjects who received at least one dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib 80 mg | Neratinib 160 mg | Neratinib 240 mg | Neratinib 320 mg
Number analyzed (Participants) | 3 | 3 | 10 | 5
Participants | 0 | 0 | 0 | 2

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of subjects who had either a complete response (CR) or partial response (PR), according to a modified Response Evaluation Criteria in Solid Tumors (RECIST). The modified RECIST is defined as CR: Disappearance of all target lesions, PR: At least a 30% decrease in the sum of the Longest Diameters (LDs) of target lesions, taking as reference the baseline sum LDs. Response required confirmation.
Time Frame: From first dose date to disease progression or last tumor assessment, up to 9.2 months
Population: Subjects who received at least 14 days of continual dose administration of drug and who had undergone at least 1 follow-up tumor assessment were considered evaluable for efficacy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib 80 mg | Neratinib 160 mg | Neratinib 240 mg | Neratinib 320 mg
Number analyzed (Participants) | 3 | 3 | 10 | 5
percentage of participants | 0 [NA to NA] — Exact Confidence Interval not computed for ORR=0% | 0 [NA to NA] — Exact Confidence Interval not computed for ORR=0% | 10.0 [0.30 to 44.5] | 20.0 [0.50 to 71.6]

3. Secondary Outcome: Clinical Benefit Rate
Description: Subjects with confirmed Complete Response (CR) or confirmed Partial Response (PR), or Stable Disease (SD) >= 24 weeks, according to a modified Response Evaluation Criteria in Solid Tumors (RECIST). SD is defined as SD in target lesions and a non-progressive disease (PD) in nontarget lesions; A PR is defined as either a PR in target lesions and a non-PD in nontarget lesions, or a CR in target lesions and an incomplete response or SD in nontarget lesions; and a CR is defined as a CR in target lesions and a CR in nontarget lesions.
Time Frame: From first dose date to progression/death or last assessment, up to 9.2 months.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib 80 mg | Neratinib 160 mg | Neratinib 240 mg | Neratinib 320 mg
Number analyzed (Participants) | 3 | 3 | 10 | 5
percentage of participants | 0 [NA to NA] — Exact Confidence Interval not computed for ORR=0% | 0 [NA to NA] — Exact Confidence Interval not computed for ORR=0% | 30.0 [6.7 to 65.2] | 40.0 [5.3 to 85.3]

4. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the prior dose level of the dose level which has >=2 of 3 to 6 subjects that experience a neratinib-related DLT during 21 days from first dose date. A DLT is defined as any HKI-272-related nonhematologic grade 3 or any grade 4 AE according to the Common Terminology Criteria for Adverse Events version 3.0 except: Grade 3 nausea, vomiting, diarrhea, or rash unless subject was receiving appropriate medical therapy.
Time Frame: First dose date through 21 days
Population: All subjects who received at least one dose.
Measure: Number; unit: mg
Arm/Group | Neratinib 240 mg
Number analyzed (Participants) | 21
mg | 240

ADVERSE EVENTS:
Time Frame: From first dose to 28 days after last dose, up to 9.2 months.
Arm/Group | Neratinib 80 mg | Neratinib 160 mg | Neratinib 240 mg | Neratinib 320 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 4/10 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 10/10 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 80 mg (N=3) | Neratinib 160 mg (N=3) | Neratinib 240 mg (N=10) | Neratinib 320 mg (N=5)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 80 mg (N=3) | Neratinib 160 mg (N=3) | Neratinib 240 mg (N=10) | Neratinib 320 mg (N=5)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 1 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 1 | 0
Trichiasis (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 4 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 10 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 4
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 2
Fatigue (General disorders) | 1 | 3 | 7 | 5
Oedema (General disorders) | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3 | 3
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Proctitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 5 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 7 | 4
Blood albumin decreased (Investigations) | 2 | 1 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 7 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2
Blood calcium decreased (Investigations) | 0 | 0 | 1 | 0
Blood calcium increased (Investigations) | 0 | 0 | 1 | 0
Blood cholesterol decreased (Investigations) | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 2 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 3
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 3
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 1
Blood glucose increased (Investigations) | 1 | 1 | 4 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 1 | 0
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 2 | 0 | 1 | 2
Blood triglycerides increased (Investigations) | 1 | 2 | 2 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 7 | 4
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 1
Monocyte count increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 1 | 1
Urine output decreased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 3 | 3
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 1
White blood cell count increased (Investigations) | 1 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Hangnail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less